CLINICAL TRIAL: NCT04973969
Title: Follicular Challenge Test to Predict Response to GnRH Agonist Triggering
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, senior physician, Assaf-Harofeh Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0304-20-ASF
Record Dates: First submitted 2021-06-13; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Other): The participants will recieve decapeptyl 0.2 mg on day 2/3 of the follicular phase.At that day, and at the day after, hormonsl profile will be documented. The hormonal profile of the day after follicular decapeptyl administration will be compared to the hormonal profile to test the predictive value.
  Interventions: Other: Decapeptyl

INTERVENTIONS:
Other: Decapeptyl — diagnosis of predictio value

SUMMARY:
GnRH agonist triggering is used during ART in order to reduce the risk of OHSS. Some studies described that in up to 5% of the cycles triggered with GnRH agonist, a lack of respone or suboptimal response was displayed.

The investigators aim to asses the possibility to predict the respone to ovulation triggering by the response to decapeptyl in the follicular phase of the same cycle.

DETAILED DESCRIPTION:
The investigators will use Decapeptyl on day 2 of menstruation followed by antagonist protocol.

Hormonal proflie including E2, P, LH, FSH will be measured. LH surge and the rest of the hormonal profile will be compared to day after ovulation triggering.

ELIGIBILITY:
Inclusion Criteria:

* patients that undergo fertility preservation

  * patients planned to freeze embryos due to PGT or surrogacy --patients at high risk for OHSS

Exclusion Criteria:

* Poor ovarian response
* known hypothalamic- pituitary dysfunction

Ages: 20 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Infertility patients
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
The response to GnRH triggering | One treatment cycle (each cycle is 28 days) for each participant (up to 28 days).
  LH levels 10-12 hours after decapeptyl trigger, number of mature oocytes

CONTACTS AND LOCATIONS:
Overall Officials: Sarit Avraham, Dr, Principal Investigator — Asaf Harofe Medical Center
Locations (1):
- Shamir medical center, Tzrifin, Israel

IPD SHARING:
Plan to Share IPD: No